CLINICAL TRIAL: NCT06690905
Title: Evaluation of the Achievement of a Pharmacodynamic Target of Piperacillin-Tazobactam for the Population With Obesity: an Open Randomized Controlled Feasibility Study
Brief Title: Evaluation of the Achievement of a Pharmacodynamic Target of Piperacillin-Tazobactam for the Population With Obesity
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: CR-CSSS Champlain-Charles-Le Moyne (Other)
Responsible Party: Principal Investigator, Benoit Crevier, Principal Investigator, CR-CSSS Champlain-Charles-Le Moyne
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-956
Record Dates: First submitted 2024-11-12; First posted 2024-11-15 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Infections; Obesity and Obesity-related Medical Conditions
Keywords: Obesity; Piperacillin-tazobactam; Pharmacodynamics
MeSH Terms: conditions — Infections; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Piperacillin-tazobactam administered in a prolonged infusion (Experimental): Piperacillin-tazobactam dose will be administered over 3 hours for piperacillin-tazobactam dosages every 6 hours or over 4 hours for piperacillin-tazobactam dosages every 8 hours.
  Interventions: Drug: Piperacillin-tazobactam administered in a prolonged infusion
- Piperacillin-tazobactam administered in a standard infusion (Active Comparator): Piperacillin-tazobactam dose will be administered over 30 minutes for every piperacilline-tazobactam administered in the study (as instructed by the drug's monograph)
  Interventions: Drug: Piperacillin-tazobactam administered in a standard infusion

INTERVENTIONS:
Drug: Piperacillin-tazobactam administered in a prolonged infusion — For patients with the prolonged infusion intervention, the piperacillin-tazobactam dose will be administered via 100 ml 0.9% NaCl mini-bags infused and a volumetric pump over 3 hours for piperacillin-tazobactam dosages every 6 hours or overs 4 hours for piperacillin-tazobactam dosages every 8 hours.
  Arms: Piperacillin-tazobactam administered in a prolonged infusion
Drug: Piperacillin-tazobactam administered in a standard infusion — For patients with the standard infusion intervention, the piperacillin-tazobactam dose will be administered over 30 minutes for every piperacilline-tazobactam administered in the study (as instructed by the drug's monograph)
  Arms: Piperacillin-tazobactam administered in a standard infusion

SUMMARY:
This study aims to evaluate the feasibility of an open randomized controlled study which would assess the proportion patients with obesity who will have a favorable pharmacodynamic parameter (i.e. fT> 100% MIC) after 24 hours of piperacillin-tazobactam administered as a prolonged intermittent infusion compared to a standard infusion.

ELIGIBILITY:
Inclusion Criteria:

* Adults (18 years and older)
* Patients hospitalized at Hôpital Charles-Le Moyne
* Obesity (as defined by a body mass index of ≥ 30 kg/m^2)
* Piperacillin-tazobactam prescription initiated within last 24 hours
* Planned duration of piperacillin-tazobactam of 24 hours or more

Exclusion Criteria:

* Documented allergy to beta-lactams of the penicillin class
* Patients with renal replacement therapy (hemodialysis, peritoneal dialysis, continuous venovenous hemodiafiltration)
* Pregnancy
* History of seizures or epilepsy, active seizures or epilepsy treated with antiepileptic drug therapy
* Patients on prolonged intermittent infusion or continuous infusion of piperacillin-tazobactam before randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2025-12-19 (Estimated)

PRIMARY OUTCOMES:
Rate of adherence to the sampling protocol | At 24 hours of treatment of piperacillin-tazobactam after randomization
  Rate of patients whose blood collection takes place 24 hours after the start of administration of piperacillin-tazobactam according to the method of administration assigned during randomization
Recruitment rate | At the randomization
  Proportion of patients meeting the eligibility criteria who consent to the study.
Achievement of a prespecified number of patients recruited per month | At the randomization
  Achievement of a number of patients recruited per month of 5 to 8 patients
Proportion of eligible patients relative to the total population who received a piperacillin-tazobactam for the study period | From the screening period to the enrollment, assessed up to 24 hours after the start of a piperacillin-tazobactam prescription
  Proportion of eligible patients relative to the total population who received a piperacilline-tazobactam for the study period

SECONDARY OUTCOMES:
Proportion of patients reaching the target of fT>MIC equal to 100% after 24 hours of piperacillin-tazobactam according to the assigned intervention | At 24 hours of treatment of piperacillin-tazobactam after randomization
  Proportion of patients reaching the target of the time the free concentration of the drug remains above the MIC during the dosing interval (i.e. fT>MIC) equal to 100% after 24 hours of piperacillin-tazobactam according to the assigned intervention
Number of days of piperacillin-tazobactam treatment under study | From enrollment to the last dose of the intervention, assessed up to 42 days
  Evaluate the number of days of piperacillin-tazobactam treatment under study
Need of escalation to carbapenems antibiotics | From enrollment to the last dose of the intervention, assessed up to 42 days
  Assess if there has been an escalation to carbapenem antibiotics
Incidence of adverse events attributed to the intervention | From enrollment to the last dose of the intervention, assessed up to 42 days
  Evaluate the incidence of adverse effects attributed to the intervention
Number of days until de-escalation to a narrower spectrum injectable antibiotic or to an oral switch | From enrollment to the last dose of the intervention, assessed up to 42 days
  Evaluate the number of days until de-escalation to a narrower spectrum injectable antibiotic or to an oral switch, if necessary

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Charles- Le Moyne, Greenfield Park, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No